CLINICAL TRIAL: NCT02388191
Title: Naproxen for Pain Control With Intrauterine Device Insertion: A Randomized Double-Blind Placebo Controlled Trial
Brief Title: Naproxen for Pain Control With Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2015P000436
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Contraception
Keywords: Contraception; Naproxen; Intrauterine devices; Pain Control
MeSH Terms: conditions — Agnosia | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen sodium (Experimental): 550 mg naproxen sodium
  Interventions: Drug: Naproxen sodium
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Drug: Naproxen sodium — 550 mg, oral, on day 1. Number of Cycles: 1
  Arms: Naproxen sodium
Other: Placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is:

1. To evaluate whether 550 mg of naproxen sodium reduces pain scores with IUD insertion on a 0-10cm visual analogue scale compared to placebo (primary outcome).
2. To evaluate whether 550 mg of naproxen sodium reduces pain scores with tenaculum placement, uterine sounding and post-procedurally on a 0-10 cm visual analog scale compared to placebo (secondary outcomes).
3. To establish if prophylactic naproxen sodium is acceptable for routine use prior to IUD insertion.

Hypothesis: The administration of naproxen sodium, 550mg orally, 1 hour prior to IUD insertion will lead to a reduction in pain scores associated with IUD insertion compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Premenopausal
* Presenting for insertion of any IUD type (i.e. Mirena, Paragard, Skyla)
* English-speaking or non-English speaking with appropriate translator available

Exclusion Criteria:

* Currently pregnant or pregnant within the last 4 weeks
* Not eligible for IUD insertion per PPLM's clinical protocols
* Presenting for IUD removal and reinsertion
* Any diagnosis of chronic pain (including fibromyalgia, endometriosis, dysmenorrhea, irritable bowel syndrome, interstitial cystitis)
* Pain medications taken within 12 hours of enrollment
* Misoprostol usage within 24 hours of enrollment
* Any known allergy or contraindication to non-steroidal anti-inflammatory drugs (including active renal disease, active hepatic disease, gastric ulcer disease or gastritis, and bleeding disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — PPLM
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ngo LL, Braaten KP, Eichen E, Fortin J, Maurer R, Goldberg AB. Naproxen Sodium for Pain Control With Intrauterine Device Insertion: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1306-1313. doi: 10.1097/AOG.0000000000001746. PMID 27824753

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Placebo tablet
Period: Overall Study
Arm/Group | Naproxen Sodium | Placebo
Started | 59 | 60
Completed | 58 | 60
Not Completed | 1 | 0
Not completed — Patient did not receive IUD | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium | Placebo | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (3.9) | 24.3 (4.2) | 23.86 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or black | 1 | 1 | 2
  White or European American | 43 | 50 | 93
  Asian | 6 | 6 | 12
  Multiracial | 3 | 2 | 5
  Other | 5 | 1 | 6
Marital status [Count of Participants; unit: Participants]
  Married | 3 | 1 | 4
  Single | 51 | 54 | 105
  Other | 4 | 5 | 9
Highest level of education [Count of Participants; unit: Participants]
  High school or high school equivalency | 5 | 4 | 9
  Some college or 2 year college | 25 | 23 | 48
  4 year college or Bachelor's degree | 23 | 22 | 45
  Graduate or professional school | 5 | 9 | 14
  Other | 0 | 2 | 2
Diagnosed with chronic pain condition (yes) [Count of Participants; unit: Participants] | 2 | 1 | 3
Diagnosed with depression (yes) [Count of Participants; unit: Participants] | 14 | 11 | 25
Baseline stress, self-report [Median (Inter-Quartile Range); unit: units on a scale] — This measure asked the following:
  "How stressed have you felt in the past week on a scale of 0-10, where 0 is not stressed at all and 10 is the most stressed ever".
  Participants were then able to circle any whole number from 0-10 to indicate their answer.
  units on a scale | 4 [3 to 6] | 4 [3 to 6] | 4 [3 to 6]
Baseline sadness, self-report [Median (Inter-Quartile Range); unit: units on a scale] — This measure asked the following:
  "How sad have you felt in the past week on a scale of 0-10, where 0 is not sad at all and 10 is the most sad ever".
  Participants were then able to circle any whole number from 0-10 to indicate their answer.
  units on a scale | 2 [1 to 3] | 3 [1 to 4] | 2 [1 to 4]
Baseline anxiety, self-report [Median (Inter-Quartile Range); unit: units on a scale] — This measure asked the following:
  "On a scale of 0 to 10, where 0 is no anxiety and 10 is the most anxious you could be, how have you been feeling in the past week?".
  Participants were then able to circle any whole number from 0-10 to indicate their answer.
  units on a scale | 3 [2 to 5] | 4 [2 to 5] | 3.5 [2 to 5]
Baseline pain tolerance, self report [Median (Inter-Quartile Range); unit: units on a scale] — This measure asked the following:
  "How would you rate your pain tolerance (ability to handle pain) in general?". Response choices included: Very low (not much at all), Low, Moderate, High, or Very High (Can tolerate a lot of pain). Patients were asked to check the box of the choice that was correct for them.
  Conversions to numerical values were as follows:
  Very low = 1 Low = 2 Moderate = 3 High = 4 Very high = 5
  units on a scale | 3 [3 to 4] | 4 [3 to 4] | 3 [3 to 4]
Expected pain for IUD insertion [Median (Inter-Quartile Range); unit: units on a scale] — This measure asked the following:
  "On a scale of 0 to 10, where 0 is no anxiety and 10 is the most anxious you could be, how anxious are you about the IUD placement?".
  Participants were then able to circle any whole number from 0-10 to indicate their answer.
  units on a scale | 45.5 [32 to 60] | 50.3 [28.8 to 62] | 49.3 [29 to 61.3]

OUTCOME MEASURES:

1. Primary Outcome: Pain at Time of IUD Insertion Using a 10 cm (100 mm) Visual Analog Scale (VAS)
Description: Pain at time of IUD insertion will be measured immediately upon completion of IUD insertion using a 100 mm visual analog scale (VAS). Patients are presented with a 100 mm line. On one end of the line, the anchor is "0 = No pain". On the opposite end of the line, the anchor is "10 = worst pain possible". Subjects are asked: "Where 0 is no pain and 10 is the worst pain possible, please record your pain on the scale below." Research staff measure the distance between the "0 = No pain" anchor and the mark made by the patient (in mm) to score the measure.
Time Frame: Immediately after IUD insertion is complete
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Naproxen Sodium | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | 69 [52.5 to 80.5] | 66 [50 to 82]

2. Secondary Outcome: Pain With Tenaculum Placement Using a 10cm (100 mm) Visual Analog Scale (VAS)
Description: Pain with tenaculum placement will be measured immediately after tenaculum is placed on the cervix using a 10cm (100 mm) visual analog scale (VAS). Patients are presented with a 100 mm line. On one end of the line, the anchor is "0 = No pain". On the opposite end of the line, the anchor is "10 = worst pain possible". Subjects are asked: "Where 0 is no pain and 10 is the worst pain possible, please record your pain on the scale below." Research staff measure the distance between the "0 = No pain" anchor and the mark made by the patient (in mm) to score the measure.
Time Frame: Immediately after tenaculum is placed on cervix
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Naproxen Sodium | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | 37.3 [20 to 55] | 31.8 [17 to 60]

3. Secondary Outcome: Pain With Uterine Sounding Using a 10cm (100 mm) Visual Analog Scale (VAS)
Description: Pain with uterine sounding will be measured immediately after uterine sounding using a 10cm (100 mm) visual analog scale (VAS). Patients are presented with a 100 mm line. On one end of the line, the anchor is "0 = No pain". On the opposite end of the line, the anchor is "10 = worst pain possible". Subjects are asked: "Where 0 is no pain and 10 is the worst pain possible, please record your pain on the scale below." Research staff measure the distance between the "0 = No pain" anchor and the mark made by the patient (in mm) to score the measure.
Time Frame: Immediately after uterine sounding
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Naproxen Sodium | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | 59.8 [45 to 75] | 58 [39 to 68]

4. Secondary Outcome: Pain 5 Minutes After IUD Insertion Using a 10cm (100 mm) Visual Analog Scale (VAS)
Description: Pain 5 minutes after IUD insertion will occur five minutes after IUD insertion is complete using a 10cm (100 mm) visual analog scale (VAS). Patients are presented with a 100 mm line. On one end of the line, the anchor is "0 = No pain". On the opposite end of the line, the anchor is "10 = worst pain possible". Subjects are asked: "Where 0 is no pain and 10 is the worst pain possible, please record your pain on the scale below." Research staff measure the distance between the "0 = No pain" anchor and the mark made by the patient (in mm) to score the measure.
Time Frame: Five minutes after IUD insertion is complete
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Naproxen Sodium | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | 16.5 [4.5 to 29] | 26 [14 to 39]

5. Secondary Outcome: Pain 15 Minutes After IUD Insertion Using a 10cm (100 mm) Visual Analog Scale (VAS)
Description: Pain 15 minutes after IUD insertion will occur 15 minutes after IUD insertion is complete using a 10cm (100 mm) visual analog scale (VAS). Patients are presented with a 100 mm line. On one end of the line, the anchor is "0 = No pain". On the opposite end of the line, the anchor is "10 = worst pain possible". Subjects are asked: "Where 0 is no pain and 10 is the worst pain possible, please record your pain on the scale below." Research staff measure the distance between the "0 = No pain" anchor and the mark made by the patient (in mm) to score the measure.
Time Frame: Fifteen minutes after IUD insertion is complete
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Naproxen Sodium | Placebo
Number analyzed (Participants) | 58 | 60
units on a scale | 12.8 [5 to 31] | 24 [11 to 38]

ADVERSE EVENTS:
Arm/Group | Naproxen Sodium | Placebo
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 2/58 | 3/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (N=58) | Placebo (N=60)
Vasovagal episode (General disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No